CLINICAL TRIAL: NCT04442048
Title: COV-IMMUNO: A Randomized, Phase III Trial of Immunization With IMM-101 Versus Observation for the Prevention of Severe Respiratory and COVID-19 Related Infections in Cancer Patients at Increased Risk of Exposure
Brief Title: Immunization With IMM-101 vs Observation for Prevention of Respiratory and Severe COVID-19 Related Infections in Cancer Patients at Increased Risk of Exposure
Acronym: COV-IMMUNO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Immodulon Therapeutics Ltd (Industry); BioCan Rx (Unknown); Canadian Cancer Society (CCS) (Other); ATGen Canada Inc (Industry); Canadian Centre for Applied Research in Cancer Control (ARCC) (Unknown); Ontario Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC8
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Covid-19
MeSH Terms: conditions — Neoplasms; COVID-19 | interventions — IMM-101; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMM-101 (Experimental): The treatment regimen with IMM-101 will be one 1.0 mg (= 0.1 mL) dose given on Day 0, followed by a second dose of 0.5 mg (= 0.05 mL) on Day 14 (-2/+5 days), and a third Dose of 0.5 mg (= 0.05 mL) on Day 45 (+/-14 days)
  Interventions: Biological: IMM-101
- Observation (Active Comparator)
  Interventions: Other: Observation

INTERVENTIONS:
Biological: IMM-101 — Three doses of IMM-101 on days 0, 14, and 45.
  Arms: IMM-101
Other: Observation — No active treatment. Observation only
  Arms: Observation

SUMMARY:
The purpose of this study is to find out if immunization with IMM-101 will reduce the incidence of severe respiratory and COVID-19 infections in cancer patients.

DETAILED DESCRIPTION:
IMM-101 is a new type of immune stimulating therapy being developed for the treatment of cancer that may also help in preventing severe respiratory and COVID-19 infections. Laboratory tests show that IMM-101 works by activating parts of the immune system that are also involved with protecting against viral and bacterial infections, so that if you are exposed to these types of infections your body may be able fight off the infection better. That could help prevent severe symptoms from respiratory and COVID-19 related infections. It has been studied in over 300 cancer patients who have also been receiving other cancer treatments, including chemotherapy and radiation, and seems promising, but it is not clear if it can offer better results than not having the immunization at all.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be undergoing (or be planned to undergo) active treatment for one or more solid malignancy, lymphoma or myeloma. active treatment includes adjuvant, neoadjuvant and palliative intent treatment with surgery, radiation, chemotherapy, targeted therapy or immunotherapy.
* Patients must have one or more of the following risk factors [CDC 2019] for a severe COVID-19 infection:

  * Age > 65 years old
  * Hypertension (on medications);
  * Type 1 or 2 Diabetes (on medication)
  * A relevant chronic condition as per the investigator based on the medical record, including:

    * heart (e.g. heart failure, coronary artery disease, congenital heart disease, cardiomyopathies, and pulmonary hypertension)
    * lung (e.g. chronic obstructive pulmonary disease (COPD including emphysema and chronic bronchitis), moderate to severe asthma, idiopathic pulmonary fibrosis and cystic fibrosis)
    * liver cirrhosis
    * serious kidney disease requiring dialysis
  * Receiving systemic therapy (such as cytotoxic chemotherapy, immunotherapy or targeted agents excluding single-agent hormonal therapy)
  * Body Mass Index > 40
  * Living in a nursing home or long term care facility
* Patient must have a life expectancy of >6 months as assessed by the investigator
* Patient must have an ECOG Performance Status ≤ 2
* Patient has adequate organ function appropriate for the therapy the patient is planned to receive in the opinion of the investigator and based on local assessment and practices.
* Patient is aged ≥ 18 years
* Patient has agreed to receive pneumococcal vaccination and a seasonal influenza vaccination in accordance with Canadian Guidelines.
* Patient is able (i.e. sufficiently fluent) and willing to complete the health utility questionnaires in either English or French.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patient must be willing to provide identifying information including provincial health insurance number to facilitate data linkage and follow up.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients enrolled on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method throughout the treatment period and for at least 3 months after discontinuation of treatment.

Exclusion Criteria:

* Patient previously received treatment with IMM-101.
* Patient cannot have either at present or in the past, a positive test for COVID-19 infection. If a patient has been tested for COVID-19, result must be confirmed as negative prior to enrollment.
* Patient cannot have experienced "flu-like symptoms" within 14 days prior to enrollment, including fever, extreme fatigue, new or worsening cough, myalgias, new or worsening dyspnea, and/or sputum production.
* Patient is receiving concomitant treatment with another investigational product or has received such treatment within the 3 weeks prior to enrollment.
* Patient has any co-existing active infection that, in the opinion of the Investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate.
* Patient has previously experienced an allergic reaction to any mycobacterial product, including the BCG vaccine.
* Patients with superficial bladder cancer or any other condition currently receiving or planned to be treated with BCG.
* Patient has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or a known history of or is known to have a positive test for Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA [qualitative]).
* Patients with prior or concurrent leukemia.
* Patient has had a prior bone marrow transplant.
* Patient is pregnant or breast-feeding
* Patient has documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents. This includes patient requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent, or depot corticosteroids in the 6 weeks before enrollment) or immunosuppressant drugs (such as azathioprine, tacrolimus, cyclosporine, etc.) within the 14 days prior to enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease. Steroids used for premedication prior to chemotherapy or as part of a chemotherapy regimen are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
The rate of "flu-like illness" which includes: | 1 year
  * WHO definition of "influenza-like illness" (ILI) [Fitzner 2018] or confirmed viral/bacterial respiratory infection AND
  * Results in a change or delay in cancer treatment or requirement for and unscheduled medical assesment, hospitalization or death.

SECONDARY OUTCOMES:
The incidence of documented COVID-19 infection (confirmed by any Health Canada approved COVID-19 test. Both symptomatic and asymptomatic infections will be documented | 1 year
The rate of severe respiratory and COVID-19 infection defined as a confirmed COVID-19 infection leading to hospitalization, ICU admission or death | 1 year
The number of events that meet the definition of the primary endpoint, as measured within the one-year follow-up (patients may meet the primary endpoint more than once and be counted multiple times). | 1 year
The incidence of COVID-19 seroconverted patients between baseline, 3 months, 6 months and 12 months | 3, 6, and 12 months
The incremental cost-effectiveness ratio (in the unit of CAD$ per life-years gained) measured with EQ-5D-5L | 1 year
Failure-free survival, as time from enrollment to recurrence or progression declared by the investigator on the basis of objective standard evaluation consistent with the disease site or death | 1 year
Overall survival (OS), as time from enrollment to death from any cause | 1 year
Incidence, frequency, and severity of AEs considered possibly, probably or definitely related to receipt of IMM-101 | 1 year
Incidence and frequency of local injection site reactions subsequent to IMM-101 administration | 1 year
Incidence and duration of ICU admission related to documented COVID-19 infection | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Auer, Study Chair — Ottawa Hospital Research Institute
Locations (8):
- Canada (8):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - CIUSSS de l'Estrie - Centre hospitalier, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No